CLINICAL TRIAL: NCT02637570
Title: Effect of Hibiscus Tea and Green Tea Supplements on Athletic Performance, Blood Pressure, Muscle Damage Indices and Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Makan Pourmasoumi, MSc Student, Food Security Research Center, Department of Community nutrition, School of Nutrition & Food Sciences, Isfahan University of Medical Sciences, Isfahan, Iran, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 394423
Record Dates: First submitted 2015-10-19; First posted 2015-12-22 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: healthy male athletes; 18-35 years old
MeSH Terms: interventions — Tea; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Hibiscus tea (Experimental): 420 mg Hibiscus 2 hour after dinner with 1 glass of cool water every day
  Interventions: Dietary Supplement: Hibiscus tea; Dietary Supplement: placebo (dextrose)
- green tea (Experimental): 450 mg green tea 2 hour after dinner with 1 glass of cool water every day
  Interventions: Dietary Supplement: green tea; Dietary Supplement: placebo (dextrose)
- control group (Placebo Comparator): 450 mg placebo (dextrose) 2 hour after dinner with 1 glass of cool water every day
  Interventions: Dietary Supplement: Hibiscus tea; Dietary Supplement: green tea

INTERVENTIONS:
Dietary Supplement: Hibiscus tea
  Arms: Hibiscus tea; control group
Dietary Supplement: green tea
  Arms: control group; green tea
Dietary Supplement: placebo (dextrose)
  Arms: Hibiscus tea; green tea

SUMMARY:
This study evaluated effect of Hibiscus tea and green tea supplements on athletic performance, blood pressure, muscle damage indices and oxidative stress in male athletes 18-35 years old and cardiovascular disease prevention approach.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 to 35 y/o
* no history of smoking or alcohol consumption
* no taking nutritional sport supplements during the last 2 months

Exclusion Criteria:

* any injury during intervention
* any inflammatory disease during the intervention

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
athletic performance assess by heart rate in step test (Harvard test). | 6 weeks
blood pressure | 6 weeks
serum's malondialdehyde | 6 weeks
  it will asses by spectrophotometry.
serum's lactate dehydrogenase | 6 weeks
  it will asses by calorimetry.

CONTACTS AND LOCATIONS:
Locations (1):
- male sports club members of Isfahan university of medical sciences, Isfahan, Iran